CLINICAL TRIAL: NCT02109237
Title: The Prevalence and Treatment of Sleep Disorders in Lung Transplant Recipients With BOS 2 & 3 and the Influence on Quality of Life and Daytime Activity.
Brief Title: Sleep Disorders in Bronchiolitis Obliterans Syndrome 2&3
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: The Prince Charles Hospital (Other Government)
Responsible Party: Principal Investigator, Anne Carle, Dr A. Fiene & Dr J Douglas, The Prince Charles Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HREC/13/QPCH/217
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Bronchiolitis Obliterans; Sleep Disordered Breathing Central
Keywords: Lung transplantation; Bronchiolitis obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bronchiolitis Obliterans 2 & 3 (Experimental): Assessment of sleep disorders and treatment if required
  Interventions: Procedure: Assessment of sleep disorders and treatment if required
- Bronchiolitis Obliterans 0 (Active Comparator): Assessment of sleep disorders and treatment if required
  Interventions: Procedure: Assessment of sleep disorders and treatment if required

INTERVENTIONS:
Procedure: Assessment of sleep disorders and treatment if required — Assessment of sleep disorders and treatment if required
  Other Names: Level 1 polysomnograpgh assessment and treatment if required

SUMMARY:
This study is to determine whether sleep disorders contribute to impaired quality of life and mobility in patients with Bronchiolitis Obliterans syndrome and whether non invasive positive airways pressure ventilation can improve sleep, quality of life and mobility in this patient group.

DETAILED DESCRIPTION:
Patients with Bronchiolitis Obliterans syndrome (BOS) 2 & 3 (25) will be matched 1:2 BOS 0 patients with similar demographics such as age, gender, BMI, time post transplant and renal dysfunction.Patients fitting inclusion/exclusion criteria once they have given informed consent will complete questionnaires on quality of life (QOL), any sleep issues they may have and be assessed by a doctor. Data from standard blood tests, respiratory function tests and physio assessments of daytime activity, mobility and muscle strength will be collected. All participants will undergo an overnight sleep study. If a sleep disorder is identified the participant will be offered appropriate treatment. All assessments with the exception of the sleep study will be repeated at 6 and 12 months post sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are post lung, heart lung and heart lung liver transplant with bronchiolitis obliterans 2 & 3
* Comparative group -Patients who are post lung, heart lung and heart lung liver transplant with bronchiolitis obliterans 0
* Identified possible sleep related disorder

Exclusion Criteria:

* Subjects who do not provide informed consent
* Subjects unable to understand the study and related procedures
* Patients with a life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
To Measure Prevalence of sleep disorders in Bronchiolitis Obliterans 2&3 patients | 12 months
  Using level one laboratory based polysomnograph

SECONDARY OUTCOMES:
Quality of life assessment using Rand SF36 standard survey | Baseline, 6 and 12 months after sleep study
  Participants will complete Rand SF36 standard survey for Quality of life. This will be completed at baseline visit and at 6 and 12 months post sleep study

OTHER OUTCOMES:
Assessment of daytime activity, mobility and muscle strength | Baseline, 6 and 12 months post sleep study
  As part of standard care transplant patients are assessed for daytime activity, mobility and muscle strength every 6months this data will be used to assess any changes post treatment for sleep disorders
Lung function assessment | Baseline, 6 and 12 months post sleep study
  Assessment of lung function to determine any variation post treatment for sleep disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Fiene, BA Med,Surg. FRACP MD, Principal Investigator — The Prince Charles Hospital; James Douglas, MBBS FRACP MD, Principal Investigator — The Prince Charles Hospital
Locations (1):
- The Prince Charles Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes